CLINICAL TRIAL: NCT05281315
Title: Cardiac Magnetic Resonance Features and Outcomes of Patients With Non-Compaction Cardiomyopathy - a Retrospective Follow-up From Pakistan
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Pirbhat Shams, Dr. Pirbhat Shams, Resident, Adult Cardiology, Department of Medicine, The Aga Khan University, Aga Khan University Hospital, Pakistan
Other Study IDs: 2020-5594-14863
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Left Ventricle Non-compaction Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients were retrospectively enrolled. This was a retrospective study and no intervention was performed. — Patients were retrospectively enrolled. This was a retrospective study and no intervention was performed.

SUMMARY:
Objective: To evaluate clinical characteristics, cardiac magnetic resonance imaging features, and outcomes of patients with left ventricle non-compaction.

DETAILED DESCRIPTION:
Left Ventricle Non-Compaction Cardiomyopathy (LVNCC) is a type of myocardial disease characterized by prominent myocardial trabeculae and recesses resulting in two distinct layers of myocardium: compacted layer and the non-compacted layer. It arises due to the failure of left ventricle (LV) maturation and compaction during intra-uterine life (1). As per the position statement from the European Society of Cardiology, LVNCC has been labelled as 'unclassified' type of cardiomyopathy. Clinical course can be complicated by heart failure, thromboembolism, or arrhythmia.

Phenotypic presentation of LVNC can range from extremely thickened layer of non-compacted myocardium to mere presence of prominent trabeculae and recesses albeit a compacted myocardium. Transthoracic echocardiography is the first tool to diagnose LVNC. However, Cardiac Magnetic Resonance (CMR) imaging has emerged as a strong tool to differentiate between LVNCC from mere hyper-trabeculated LV myocardium when echocardiogram is inconclusive (Figure 1 and Video 1). Various criteria have evolved to diagnose LVNC by CMR. Peterson et al defined the end-diastole non-compacted to compacted myocardium ratio of >2.3 to have good sensitivity, specificity, and negative predictive value for differentiating pathological non-compaction from hyper-trabeculation.

With an increase in the use of diagnostic cardiovascular imaging modalities in South-Asian (SA) belt, LVNC is being increasingly diagnosed. The exact prevalence of LVNC in SA is not known and phenotypic CMR characteristics, clinical features, and outcomes of LVNC remain unknown for SA population. This brought us to the need of analysing CMR data of LVNC at our centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years, referred for CMR for further evaluation of cardiomyopathy.

Exclusion Criteria:

* patients with intracardiac masses, pericardial diseases and congenital heart diseases were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively enrolled 294 patients referred for CMR from 2011 to 2020 for evaluation of cardiomyopathy. Of these, 51% were ischemic cardiomyopathy, 26% were dilated cardiomyopathy, 25% were hypertrophic cardiomyopathy, 13% were restrictive cardiomyopathy, and 6% were arrhythmogenic right ventricle dysplasia. For final enrolment, patients with intracardiac masses, pericardial diseases and congenital heart diseases were excluded from the study. Patients with evidence of LV non-compaction were further analysed for baseline characteristics, CMR parameters and outcomes. Characteristics of this group were compared with 47 patients who had dilated cardiomyopathy without evidence of LV non-compaction.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical characteristics, cardiac magnetic resonance imaging features, and outcomes of patients with left ventricle non-compaction. | 37 months
  Evaluating CMR features and looking at outcomes such as all cause mortality, major heart failure or arrhythmia hospitalizations.

SECONDARY OUTCOMES:
All cause-mortality, heart failure hospitalization, and arrhythmia hospitalization. | 37 months
  All cause-mortality, heart failure hospitalization, and arrhythmia hospitalization.

IPD SHARING:
Plan to Share IPD: No